CLINICAL TRIAL: NCT03492801
Title: Longitudinal Monitoring of Tumor Specific Mutations in Patients With Lung Cancer
Brief Title: Collection of Blood Samples in Patients With Non-small Cell Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2L-17-1; NCI-2017-02277 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2L-17-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-03-27; First posted 2018-04-10 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Stage III Non-Small Cell Lung Cancer AJCC v7; Stage IIIA Non-Small Cell Lung Cancer AJCC v7; Stage IIIB Non-Small Cell Lung Cancer AJCC v7; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection): Patients undergo collection of blood samples at baseline and every 12 weeks for up to 6 times.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot research trial studies the collection of blood samples in monitoring tumor specific mutations in patients with non-small cell lung cancer that has spread to other places in the body or cannot be removed by surgery. Collecting blood samples may help measure the changes in lung cancer, better learn methods to track cancer in the bloodstream, and improve cancer treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the ability of next generation sequencing (NGS) to monitor the evolution of cancer-specific mutations in patients undergoing treatment for non-small cell lung carcinoma and for whom the molecular profile of the tumor cells prior to treatment is known.

II. Compare the sensitivity of digital droplet polymerase chain reaction (ddPCR) to that of NGS for detecting the appearance of EGFR T790M mutations in patients treated with an EGFR tyrosine kinase inhibitor.

OUTLINE:

Patients undergo collection of blood samples at baseline and every 12 weeks for up to 6 times.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of non-small cell lung carcinoma for which the molecular profile of the primary tumor has been obtained from a block of paraffin-embedded, formalin-fixed tissue that remains available
* Zubrod performance status 0 or 1
* Patients must have metastatic or unresectable disease and be starting a new line of systemic treatment at the time of enrollment; there are no constraints regarding the time interval between the initial collection of samples for molecular profiling studies at the time of diagnosis prior to treatment and subsequent collections of circulating cell-free deoxyribonucleic acid (DNA) or circulating tumor cells
* Patients must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* Ability to understand and the willingness to sign a written informed consent; Note: There will be no discrimination between type of treatment or whether they are on continuous versus intermittent therapy

Exclusion Criteria:

* Known severe anemia (hemoglobin [Hb] < 8g/dL)
* Patients will be excluded if trackable driver mutations are not identified in the primary tumor tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are seen at all the USC facilities who have metastatic or unresectable non-small cell lung carcinoma and will be starting a new line of systemic treatment will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Blood sample collection for tumor specific mutations study from patients with non-small cell lung cancer | Baseline to 3 years
  Blood samples collected will be used to evaluate the ability of next generation sequencing (NGS) to monitor the evolution of cancer-specific mutations in patients undergoing treatment for non-small cell lung carcinoma and for whom the molecular profile of the tumor cells prior to treatment is known.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Ward, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States